CLINICAL TRIAL: NCT01806688
Title: A Randomized, Controlled, Cross-over Study of the Effect of Snacks on Appetite Control
Brief Title: Effect of Snacks on Appetite Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: Manitoba Agri-Health Research Network (Other)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principal Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H2013:036; RRC/2013/1276 (Other: Research Review Committee)
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Healthy Canadians; Appetite Control
Keywords: satiety; appetite; snack

STUDY DESIGN:
Intervention Model Description: Randomized crossover
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Snack #1 (Experimental): One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #1 is a gluten-free high protein snack comprised of a 30g serving of buckwheat groats. The placebo comparator reference product is a gluten-free snack with similar energy density, but 1/2 the protein as snack #1, comprised of a 32g serving of corn nuts. The placebo comparator non-caloric control is water.
  Interventions: Other: gluten-free high protein snack #1; Other: gluten-free snack with similar energy density but 1/2 the protein as snack #1; Other: non-caloric control
- Experimental Snack #2 (Experimental): One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #2 is a gluten-free high protein and high fibre snack comprised of a 50g serving of a buckwheat and pinto bean flour pita bread. The placebo comparator reference product is a gluten-free snack with similar energy density, but less protein and fibre than snack #2, comprised of a 50g serving of rice bread. The placebo comparator non-caloric control is water.
  Interventions: Other: non-caloric control; Other: gluten-free high protein and high fibre snack #2; Other: gluten-free snack with similar energy density, but less protein and fibre than snack #2

INTERVENTIONS:
Other: gluten-free high protein snack #1 — buckwheat groats 30g serving
  Arms: Experimental Snack #1
Other: gluten-free snack with similar energy density but 1/2 the protein as snack #1 — 32g serving of corn nuts
  Arms: Experimental Snack #1
Other: non-caloric control — water
Other: gluten-free high protein and high fibre snack #2 — buckwheat and pinto bean flour pita bread 50g serving
  Arms: Experimental Snack #2
Other: gluten-free snack with similar energy density, but less protein and fibre than snack #2 — 50g serving of rice bread
  Arms: Experimental Snack #2

SUMMARY:
This clinical trial is being conducted to study whether eating certain snacks will reduce your desire to eat and for a longer period of time compared to other snacks. The investigators are testing 2 different snacks. Study #1 will involve eating 2 different seed-like snacks or water. Study #2 will involve eating pita bread with jam, bread with jam or water. The test snack is higher in protein and/or fibre compared to the reference product.

DETAILED DESCRIPTION:
Healthy adults will be recruited to participate in a randomized, controlled, crossover study to investigate whether or not eating snacks made with buckwheat would increase satiety and reduce their energy intake when compared to a comparable snack. Water was included as a non-caloric control. The study consisted of 3 visits and participants would receive a different treatment at each visit. Visits were scheduled at least 7 days apart. Visual analog scales will be used to assess appetite related sensations at 7 time points, fasting, 30 minutes after consuming the snack and then at 30 minute intervals for 180 minutes. Participants will be provided with a lunch and the amount of food consumed will be weighed. I addition, participants will be asked to maintain a food record for the remainder of the day.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18-30kg/m2
* males and non-pregnant or non-lactating females

Exclusion Criteria:

* Diagnosis of disease by a medical doctor that requires medical treatment during the study period.
* Daily tobacco use.
* Physical Activity Level >1.8.
* Eat meals at irregular or unusual times.
* Food allergy, aversion or unwillingness to eat study foods.
* Use of any prescription or non-prescription drug, herbal or nutritional supplement known to affect appetite.
* Presence of a gastrointestinal disorder.
* Score >65% on any 1 of the 3 categories of the Three Factor Eating Questionnaire-R18.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-07-06 (Actual); Primary Completion 2014-08-23 (Actual); Study Completion 2014-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Blewett, PhD, Principal Investigator — St. Boniface Hospital Research Centre
Locations (1):
- I. H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Group results will be emailed or mailed to individuals upon request once they are available.

REFERENCES:
- [Background] Blundell J, de Graaf C, Hulshof T, Jebb S, Livingstone B, Lluch A, Mela D, Salah S, Schuring E, van der Knaap H, Westerterp M. Appetite control: methodological aspects of the evaluation of foods. Obes Rev. 2010 Mar;11(3):251-70. doi: 10.1111/j.1467-789X.2010.00714.x. Epub 2010 Jan 29. PMID 20122136
- [Background] Paddon-Jones D, Westman E, Mattes RD, Wolfe RR, Astrup A, Westerterp-Plantenga M. Protein, weight management, and satiety. Am J Clin Nutr. 2008 May;87(5):1558S-1561S. doi: 10.1093/ajcn/87.5.1558S. PMID 18469287
- [Background] Belski R. Fiber, protein, and lupin-enriched foods: role for improving cardiovascular health. Adv Food Nutr Res. 2012;66:147-215. doi: 10.1016/B978-0-12-394597-6.00004-5. PMID 22909980
- See also: Obesity in Canada: A joint report from the Public Health Agency of Canada and the Canadian Institute for Health Information — http://www.phac-aspc.gc.ca/hp-ps/hl-mvs/oic-oac/assets/pdf/oic-oac-eng.pdf
- See also: Draft guidance document: Satiety health claims on food from Health Canada — http://www.hc-sc.gc.ca/fn-an/consult/satiety-satiete/document-consultation-eng.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 289 candidates were screened between June 2013 and August 2014. Of these 289 candidates, 50 met the criteria and were determined to be eligible. The first participant was enrolled on July 6, 2013 and the last participant enrolled August 9, 2014. 46 participants were enrolled in the overall study and 30 of these completed both the seed study and the pita study while 16 participated in only one of the studies. 38 participants were randomized to the seed study and 38 to the pita study.
Pre-assignment Details: 30 people completed both studies and 16 participated in only 1 study.
Groups:
- Seed Study: One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #1 is a gluten-free high protein snack comprised of a 30g serving of buckwheat groats. The placebo comparator reference product is a gluten-free snack with similar energy density, but 1/2 the protein as snack #1, comprised of a 32g serving of corn nuts. The placebo comparator non-caloric control is water.
- Pita Study: One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #2 is a gluten-free high protein and high fibre snack comprised of a 50g serving of a buckwheat and pinto bean flour pita bread. The placebo comparator reference product is a gluten-free snack with similar energy density, but less protein and fibre than snack #2, comprised of a 50g serving of rice bread. The placebo comparator non-caloric control is water.
Period: First Intervention Seed Study
Arm/Group | Seed Study | Pita Study
Started (Day 1) | 38 (Participants received one of the following: 1. experimental snack #1 gluten-free high protein snack a 30 g serving of buckwheat groats 2. placebo comparator reference product, a gluten-free snack with similar energy density but 1/2 the protein as the experimental snack, a 32g serving of corn nuts 3. placebo comparator non-caloric control water) | 0 (Participants received one of the following: 1. experimental snack #1 gluten-free high protein snack a 30 g serving of buckwheat groats 2. placebo comparator reference product, a gluten-free snack with similar energy density but 1/2 the protein as the experimental snack, a 32g serving of corn nuts 3. placebo comparator non-caloric control water)
Experimental Snack #1 | 13 (Received experimental snack #1 at the first visit, a 30g serving of buckwheat groats) | 0 (Received experimental snack #1 at the first visit, a 30g serving of buckwheat groats)
Placebo Comparator Reference Product #1 | 13 (Received the placebo comparator reference product #1 at the first visit, a 32g serving of corn nuts) | 0 (Received the placebo comparator reference product #1 at the first visit, a 32g serving of corn nuts)
Placebo Comparator Non-caloric Control #1 | 12 (Received water, the placebo comparator non-caloric control #1 at the first visit) | 0 (Received water, the placebo comparator non-caloric control #1 at the first visit)
Completed | 38 | 0
Not Completed | 0 | 0
Period: Second Intervention Seed Study
Arm/Group | Seed Study | Pita Study
Started (Day 8) | 38 (Participants received one of the following they hadn't previously received at visit 1: 1. experimental snack #1 gluten-free high protein snack a 30 g serving of buckwheat groats 2. placebo comparator reference product #1, a gluten-free snack with similar energy density but 1/2 the protein as the experimental snack, a 32g serving of corn nuts 3. placebo comparator non-caloric control #1, water) | 0 (Participants received one of the following they hadn't previously received at visit 1: 1. experimental snack #1 gluten-free high protein snack a 30 g serving of buckwheat groats 2. placebo comparator reference product #1, a gluten-free snack with similar energy density but 1/2 the protein as the experimental snack, a 32g serving of corn nuts 3. placebo comparator non-caloric control #1, water)
Experimental Snack #1 | 13 (Received the experimental snack #1, a 30g serving of buckwheat groats at visit 2) | 0 (Received the experimental snack #1, a 30g serving of buckwheat groats at visit 2)
Placebo Comparator Reference Product #1 | 13 (Received the Placebo comparator reference product #1, a 32g serving of corn nuts at visit 2) | 0 (Received the Placebo comparator reference product #1, a 32g serving of corn nuts at visit 2)
Placebo Comparator Non-caloric Control #1 | 12 (Received water, the placebo comparator non-caloric control #1 at visit 2) | 0 (Received water, the placebo comparator non-caloric control #1 at visit 2)
Completed | 38 | 0
Not Completed | 0 | 0
Period: Third Intervention Seed Study
Arm/Group | Seed Study | Pita Study
Started (Day 15) | 38 (Participants received one of the following they hadn't previously received at visit 1 or visit 2: 1. experimental snack #1 gluten-free high protein snack a 30 g serving of buckwheat groats 2. placebo comparator reference product, a gluten-free snack with similar energy density but 1/2 the protein as the experimental snack, a 32g serving of corn nuts 3. placebo comparator non-caloric control water) | 0 (Participants received one of the following they hadn't previously received at visit 1 or visit 2: 1. experimental snack #1 gluten-free high protein snack a 30 g serving of buckwheat groats 2. placebo comparator reference product, a gluten-free snack with similar energy density but 1/2 the protein as the experimental snack, a 32g serving of corn nuts 3. placebo comparator non-caloric control water)
Experimental Snack #1 | 12 (Received the Experimental snack #1, a 30g serving of buckwheat groats at visit 3) | 0 (Received the Experimental snack #1, a 30g serving of buckwheat groats at visit 3)
Placebo Comparator Reference Product #1 | 12 (Received the placebo comparator reference product #1, a 32g serving of corn nuts at visit 3) | 0 (Received the placebo comparator reference product #1, a 32g serving of corn nuts at visit 3)
Placebo Comparator Non-caloric Control #1 | 14 (Received water, the placebo comparator non-caloric control #1 at visit 3) | 0 (Received water, the placebo comparator non-caloric control #1 at visit 3)
Completed | 38 | 0
Not Completed | 0 | 0
Period: First Intervention Pita Study
Arm/Group | Seed Study | Pita Study
Started (Day 1) | 0 (Participants received one of the following: 1. experimental snack #2 gluten-free high protein and high fibre snack a 50 g serving of buckwheat and pinto bean flour pita bread 2. placebo comparator reference product, a gluten-free snack with similar energy density but less protein and fibre as the experimental snack, a 50g serving of rice bread 3. placebo comparator non-caloric control water) | 38 (Participants received one of the following: 1. experimental snack #2 gluten-free high protein and high fibre snack a 50 g serving of buckwheat and pinto bean flour pita bread 2. placebo comparator reference product, a gluten-free snack with similar energy density but less protein and fibre as the experimental snack, a 50g serving of rice bread 3. placebo comparator non-caloric control water)
Experimental Snack #2 | 0 (Received the Experimental snack #2, a 50 g serving of buckwheat and pinto bean flour pita bread at the first visit) | 14 (Received the Experimental snack #2, a 50 g serving of buckwheat and pinto bean flour pita bread at the first visit)
Placebo Comparator Reference Product #2 | 0 (Received the placebo comparator reference product #2 at the first visit, a 50g serving of rice bread) | 12 (Received the placebo comparator reference product #2 at the first visit, a 50g serving of rice bread)
Placebo Comparator Non-caloric Control #2 | 0 (Received water, the placebo comparator non-caloric control #2 at the first visit) | 12 (Received water, the placebo comparator non-caloric control #2 at the first visit)
Completed | 0 | 38
Not Completed | 0 | 0
Period: Second Intervention Pita Study
Arm/Group | Seed Study | Pita Study
Started (Day 8) | 0 (Participants received one of the following: 1. experimental snack #2 gluten-free high protein and high fibre snack a 50 g serving of buckwheat and pinto bean flour pita bread 2. placebo comparator reference product, a gluten-free snack with similar energy density but less protein and fibre as the experimental snack, a 50g serving of rice bread 3. placebo comparator non-caloric control water) | 38 (Participants received one of the following: 1. experimental snack #2 gluten-free high protein and high fibre snack a 50 g serving of buckwheat and pinto bean flour pita bread 2. placebo comparator reference product, a gluten-free snack with similar energy density but less protein and fibre as the experimental snack, a 50g serving of rice bread 3. placebo comparator non-caloric control water)
Experimental Snack #2 | 0 (Received the Experimental snack #2, a 50 g serving of buckwheat and pinto bean flour pita bread at the second visit) | 12 (Received the Experimental snack #2, a 50 g serving of buckwheat and pinto bean flour pita bread at the second visit)
Placebo Comparator Reference Product #2 | 0 (Received the placebo comparator reference product #2 at the second visit, a 50g serving of rice bread) | 13 (Received the placebo comparator reference product #2 at the second visit, a 50g serving of rice bread)
Placebo Comparator Non-caloric Control #2 | 0 (Received water, the placebo comparator non-caloric control #2 at the second visit) | 13 (Received water, the placebo comparator non-caloric control #2 at the second visit)
Completed | 0 | 38
Not Completed | 0 | 0
Period: Third Intervention Pita Study
Arm/Group | Seed Study | Pita Study
Started (Day 15) | 0 (Participants received one of the following: experimental snack #2 gluten-free high protein and high fibre snack a 50 g serving of buckwheat and pinto bean flour pita bread placebo comparator reference product, a gluten-free snack with similar energy density but less protein and fibre as the experimental snack, a 50g serving of rice bread placebo comparator non-caloric control water) | 38 (Participants received one of the following: experimental snack #2 gluten-free high protein and high fibre snack a 50 g serving of buckwheat and pinto bean flour pita bread placebo comparator reference product, a gluten-free snack with similar energy density but less protein and fibre as the experimental snack, a 50g serving of rice bread placebo comparator non-caloric control water)
Experimental Snack #2 | 0 (Received the Experimental snack #2, a 50 g serving of buckwheat and pinto bean flour pita bread at the third visit) | 12 (Received the Experimental snack #2, a 50 g serving of buckwheat and pinto bean flour pita bread at the third visit)
Placebo Comparator Reference Product #2 | 0 (Received the placebo comparator reference product #2 at the third visit, a 50g serving of rice bread) | 13 (Received the placebo comparator reference product #2 at the third visit, a 50g serving of rice bread)
Placebo Comparator Non-caloric Control #2 | 0 (Received water, the placebo comparator non-caloric control #2 at the third visit) | 13 (Received water, the placebo comparator non-caloric control #2 at the third visit)
Completed | 0 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There are two arms to this study, the Seed Study and the Pita Study. A total of 46 participants were enrolled in the overall study, and of those 46 enrolled, 30 people participated in both studies while 16 only participated in one study. 38 participants were randomized to complete the Seed Study and 38 participants were randomized to complete the Pita Study.
Groups:
- Pita Study: One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #2 is a gluten-free high protein and high fibre snack comprised of a 50g serving of buckwheat and pinto bean flour pita bread. The placebo comparator reference product is a gluten-free snack with similar energy density, but less protein and fibre than snack #2, comprised of a 50g serving of rice bread. The placebo comparator non-caloric control is water.
- Total: Total of all reporting groups
Arm/Group | Seed Study | Pita Study | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants] — Population: 289 candidates were screened for the study between June 2013 and August 2014. Of those 289 candidates, 50 met the inclusion criteria and of those 50, a total of 46 were enrolled in the overall study. 38 were randomized to treatment in the Seed Study and 38 were randomized to treatment in the Pita Study. 30 completed both studies and 16 chose to do just one study.
  Participants
    Seed Study: number analyzed (Participants) | 38 | 0 | 38
    Seed Study: <=18 years | 0 | 0 | 0
    Seed Study: Between 18 and 65 years | 37 | 0 | 37
    Seed Study: >=65 years | 1 | 0 | 1
    Pita Study: number analyzed (Participants) | 0 | 38 | 38
    Pita Study: <=18 years | 0 | 0 | 0
    Pita Study: Between 18 and 65 years | 0 | 37 | 37
    Pita Study: >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] — Population: A total of 46 participants were enrolled in the overall study, and of those 46 enrolled, 30 participated in both studies while 16 only participated in one study. 38 participants were randomized to complete the Seed Study and 38 participants to complete the Pita Study.
  years
    Seed Study: number analyzed (Participants) | 38 | 0 | 38
    Seed Study | 37.7 [20 to 67] |  | 37.7 [20 to 67]
    Pita Study: number analyzed (Participants) | 0 | 38 | 38
    Pita Study |  | 33.5 [20 to 67] | 33.5 [20 to 67]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 46 participants were enrolled in the overall study, and of those 46 enrolled, 30 participated in both studies while 16 only participated in one study. 38 participants were randomized to complete the Seed Study and 38 participants to complete the Pita Study.
  Participants
    Seed Study: number analyzed (Participants) | 38 | 0 | 38
    Seed Study: Female | 10 | 0 | 10
    Seed Study: Male | 28 | 0 | 28
    Pita Study: number analyzed (Participants) | 0 | 38 | 38
    Pita Study: Female | 0 | 11 | 11
    Pita Study: Male | 0 | 27 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 46 participants were enrolled in the overall study, and of those 46 enrolled, 30 participated in both studies while 16 only participated in one study. 38 participants were randomized to complete the Seed Study and 38 participants to complete the Pita Study.
  Participants
    Seed Study: number analyzed (Participants) | 38 | 0 | 38
    Seed Study: American Indian or Alaska Native | 0 | 0 | 0
    Seed Study: Asian | 9 | 0 | 9
    Seed Study: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Seed Study: Black or African American | 0 | 0 | 0
    Seed Study: White | 24 | 0 | 24
    Seed Study: More than one race | 2 | 0 | 2
    Seed Study: Unknown or Not Reported | 3 | 0 | 3
    Pita Study: number analyzed (Participants) | 0 | 38 | 38
    Pita Study: American Indian or Alaska Native |  | 0 | 0
    Pita Study: Asian |  | 11 | 11
    Pita Study: Native Hawaiian or Other Pacific Islander |  | 0 | 0
    Pita Study: Black or African American |  | 1 | 1
    Pita Study: White |  | 20 | 20
    Pita Study: More than one race |  | 3 | 3
    Pita Study: Unknown or Not Reported |  | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants] — Seed Study Population: Data collected from the two studies are reported in separate Baseline Measures
  Participants
    Canada: number analyzed (Participants) | 38 | 0 | 38
    Canada | 38 | 0 | 38
Region of Enrollment [Count of Participants; unit: Participants] — Pita Study Population: Data collected from the two studies are reported in separate Baseline Measures
  Participants
    Canada: number analyzed (Participants) | 0 | 38 | 38
    Canada | 0 | 38 | 38

OUTCOME MEASURES:

1. Primary Outcome: Total Area Under the Curve (AUC) for Hunger, Fullness, Desire to Eat and Prospective Consumption Using Visual Analog Scales (VAS)
Description: Appetite assessment was measured using a VAS questionnaire administered pre-snack and every 30 minutes post snack up to 180 minutes, for a total of 7 time points. The questionnaire included 4 questions (1) How hungry are you? (2) How full are you? (3) How strong is your desire to eat? (4) How much do you think you want to eat right now? Each question was followed by a 10 cm line anchored at the left and right ends by the opposing statements "not at all" and "extremely" for questions 1 and 2, "very weak " and "very strong" for question 3, and "nothing at all" and "a very large amount" for question 4. Participants provided their response to each question by marking a perpendicular line on the 10-cm line to indicate their answer. Scores were determined by measuring the distance in centimeters from the left anchor to the perpendicular line drawn by the participant. VAS scores over time were graphed and AUC was calculated using the trapezoid method.
Time Frame: VAS administered pre-snack and then every 30 minutes after the first bite up to 180 minutes for a total of 7 time points.
Population: A total of 46 participants were enrolled in the Seed and the Pita Study. Of these 46, 30 participated in both studies and 16 enrolled in just one study. 38 participants enrolled in the Seed Study and 38 in the Pita Study.
Measure: Least Squares Mean (Standard Error); unit: cm x min
Groups:
- Pita Study: One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #2 is a gluten-free high protein and high fibre snack comprised of a 50g serving of buckwheat and pinto bean flour pita bread. The placebo comparator reference product is a gluten-free snack with similar energy density but less protein and fiber than snack #2, comprised of a 50g serving of rice bread. The placebo comparator non-caloric control is water.
Arm/Group | Seed Study | Pita Study
Number analyzed (Participants) | 37 | 37
cm x min
  Seed Study Experimental Snack #1 Hunger: number analyzed (Participants) | 37 | 0
  Seed Study Experimental Snack #1 Hunger | 651 (46) |
  Seed Study Experimental Snack #1 Fullness: number analyzed (Participants) | 37 | 0
  Seed Study Experimental Snack #1 Fullness | 1008 (46) |
  Seed Study Experimental Snack #1 Desire: number analyzed (Participants) | 37 | 0
  Seed Study Experimental Snack #1 Desire | 638 (46) |
  Seed Study Experimental Snack #1 Consume: number analyzed (Participants) | 37 | 0
  Seed Study Experimental Snack #1 Consume | 640 (42) |
  Seed Study Placebo Comparator #1 Hunger: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Comparator #1 Hunger | 636 (46) |
  Seed Study Placebo Comparator #1 Fullness: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Comparator #1 Fullness | 1024 (46) |
  Seed Study Placebo Comparator #1 Desire: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Comparator #1 Desire | 659 (46) |
  Seed Study Placebo Comparator #1 Consume: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Comparator #1 Consume | 649 (42) |
  Seed Study Placebo Comparator #1 Non-caloric Control Hunger: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Comparator #1 Non-caloric Control Hunger | 962 (46) |
  Seed Study Placebo Control #1 Non-caloric Control Fullness: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Control #1 Non-caloric Control Fullness | 682 (47) |
  Seed Study Placebo Control #1 Non-caloric Control Desire: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Control #1 Non-caloric Control Desire | 980 (47) |
  Seed Study Placebo Comparator Non-caloric Control #1 Consume: number analyzed (Participants) | 37 | 0
  Seed Study Placebo Comparator Non-caloric Control #1 Consume | 916 (42) |
  Pita Study Experimental Snack #2 Hunger: number analyzed (Participants) | 0 | 37
  Pita Study Experimental Snack #2 Hunger |  | 611 (40)
  Pita Study Experimental Snack #2 Fullness: number analyzed (Participants) | 0 | 37
  Pita Study Experimental Snack #2 Fullness |  | 1005 (41)
  Pita Study Experimental Snack #2 Desire: number analyzed (Participants) | 0 | 37
  Pita Study Experimental Snack #2 Desire |  | 616 (44)
  Pita Study Experimental Snack #2 Consume: number analyzed (Participants) | 0 | 37
  Pita Study Experimental Snack #2 Consume |  | 599 (38)
  Pita Study Placebo Comparator #2 Reference Product Hunger: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Reference Product Hunger |  | 661 (39)
  Pita Study Placebo Comparator #2 Reference Product Fullness: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Reference Product Fullness |  | 968 (40)
  Pita Study Placebo Comparator #2 Reference Product Desire: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Reference Product Desire |  | 682 (43)
  Pita Study Placebo Comparator #2 Reference Product Consume: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Reference Product Consume |  | 676 (38)
  Pita Study Placebo Comparator #2 Non-caloric Control Hunger: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Non-caloric Control Hunger |  | 956 (39)
  Pita Study Placebo Comparator #2 Non-caloric Control Fullness: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Non-caloric Control Fullness |  | 675 (40)
  Pita Study Placebo Comparator #2 Non-caloric Control Desire: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Non-caloric Control Desire |  | 1001 (43)
  Pita Study Placebo Comparator #2 Non-caloric Control Consume: number analyzed (Participants) | 0 | 37
  Pita Study Placebo Comparator #2 Non-caloric Control Consume |  | 959 (38)
Statistical Analysis 1: Comparison: Seed Study vs Pita Study; Items #1 were compared to each other and Items #2 were compared to each other; Test type: Equivalence — The study is designed to detect a 10.0% difference in area under the curve (AUC) appetite ratings between foods. The required number of Participants is 38; p < 0.05, ANCOVA; Sources of variation included in the model: snack, visit number, baseline score, visit number × snack, and snack × overweight

2. Secondary Outcome: Number of Calories Consumed Post-snack Until Bedtime
Description: Participants were provided with a food diary to record the amount and type of each food and beverage consumed for the remainder of the day. Energy consumed at lunch and the remainder of the day were quantified from food consumed at lunch and the food diary using Food Processor Nutrient Analysis Software.
Time Frame: time between snack consumption and bedtime (12 hours)
Population: In the Seed Study data for 36 participants was analyzed. One participant was not analyzed due to non compliance and a second participant for not providing a food record. In the Pita Study data from 34 participants was analyzed. One participant was noncompliant and 3 did not turn in food records.
Measure: Mean (Standard Error); unit: kcal
Groups:
- Pita Study: One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #2 is a gluten-free high protein and high fibre snack comprised of a 50g serving of buckwheat pita. The placebo comparator reference product is a gluten-free snack with similar energy density, but less protein and fibre than snack #2, comprised of a 50g serving of rice bread. The placebo comparator non-caloric control is water.
Arm/Group | Seed Study | Pita Study
Number analyzed (Participants) | 36 | 34
kcal
  Seed Study Experimental Snack #1: number analyzed (Participants) | 36 | 0
  Seed Study Experimental Snack #1 | 1429 (70) |
  Seed Study Placebo Comparator #1 Reference Product: number analyzed (Participants) | 36 | 0
  Seed Study Placebo Comparator #1 Reference Product | 1326 (94) |
  Seed Study Placebo Comparator #1 Non-caloric Control: number analyzed (Participants) | 36 | 0
  Seed Study Placebo Comparator #1 Non-caloric Control | 1288 (80) |
  Pita Study Experimental Snack #2: number analyzed (Participants) | 0 | 34
  Pita Study Experimental Snack #2 |  | 1448 (89)
  Pita Study Placebo Comparator #2 Reference Product: number analyzed (Participants) | 0 | 34
  Pita Study Placebo Comparator #2 Reference Product |  | 1414 (78)
  Pita Study Placebo Comparator #2 Non-caloric Control: number analyzed (Participants) | 0 | 34
  Pita Study Placebo Comparator #2 Non-caloric Control |  | 1478 (75)
Statistical Analysis 1: Comparison: Seed Study; Items #1 were compared to each other and Items #2 were compared to each other; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Gastrointestinal Side Effects
Description: Participants were asked if they noticed any gastrointestinal side effects after having eaten the study food and the results were recorded.
Time Frame: 24h
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Likeability of Test and Reference Products Based on Sensory Scales
Description: Likability of the study products was assessed using a 5-point hedonic scale (1 = dislike extremely; 2 = dislike very moderately; 3 = neither like or dislike; 4 = like moderately; 5 = like extremely) for appearance, aroma, flavour, taste, texture and overall liking.
Time Frame: immediately after eating test or reference product
Measure: Least Squares Mean (Standard Error); unit: sensory rating on a scale of 1 to 5
Groups:
- Experimental Snack #2: One of three interventions to be administered at each visit, an experimental snack, a placebo comparator reference product or a placebo comparator non-caloric control. The experimental snack #2 is a gluten-free high protein and high fibre snack comprised of a 50g serving of buckwheat and pinto bean flour pita bread. The placebo comparator reference product is a gluten-free snack with similar energy density, but less protein and fibre than snack #2, comprised of a 50g serving of rice bread. The placebo comparator non-caloric control is water.
Arm/Group | Experimental Snack #1 | Experimental Snack #2
Number analyzed (Participants) | 38 | 38
sensory rating on a scale of 1 to 5
  Experimental Snack taste | 3.57 (.2) | 3.66 (.15)
  Experimental Snack texture | 3.66 (.19) | 3.49 (.19)
  Experimental Snack appearance | 3.57 (.16) | 3.81 (.14)
  Experimental Snack overall | 3.48 (.18) | 3.64 (.15)
  Experimental Snack aroma | 3.4 (.11) | 3.45 (.10)
  Placebo Comparator Reference taste | 3.23 (.20) | 3.67 (.15)
  Placebo Comparator Reference texture | 2.64 (.19) | 3.36 (.19)
  Placebo Comparator Reference appearance | 3.49 (.16) | 3.74 (.14)
  Placebo Comparator Reference aroma | 3.34 (.11) | 3.39 (.10)
  Placebo Comparator Reference overall | 3.05 (.18) | 3.58 (.14)
Statistical Analysis 1: Comparison: Experimental Snack #1; Items #1 were compared to each other and Items #2 were compared to each other; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: No adverse events.
Arm/Group | Seed Study | Pita Study
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No